CLINICAL TRIAL: NCT00285792
Title: Stanford Preschool Physical Activity Project
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 96534
Record Dates: First submitted 2006-01-31; First posted 2006-02-02 (Estimated); Last update posted 2006-10-05 (Estimated); Status verified 2006-07

CONDITIONS: Obesity
Keywords: Preschool, Physical Activity
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Exercise

INTERVENTIONS:
Behavioral: Physical Activity

SUMMARY:
The purpose of this study is to examine the effects of increasing the amount of time spent in recess (outside playtime) on overall daily physical activity in Hispanic preschool age children attending full-day and half-day preschool programs. We hypothesize that increasing recess (outside playtime) by 60 minutes in participants attending full-day and 30 minutes in participants attending half-day of preschool will increase average daily physical activity during the intervention days. We also hypothesize that children will not compensate for the increased recess (outside playtime) by decreasing physical activity outside of school during the intervention days.

DETAILED DESCRIPTION:
Childhood obesity has dramatically increased in the past two decades. The increased prevalence of obesity in Hispanic children is even more alarming. Obesity is a known risk factor for the development of a wide range of chronic diseases in both children and adults, and overweight status tends to track from childhood into adulthood. Therefore, many experts have recommended that obesity prevention should be initiated during early childhood, particularly in preschool-aged children, to prevent the excess co-morbidities associated with obesity throughout the lifespan. However, less is known about the prevention of obesity in young children.

One factor associated with the increased prevalence of overweight and obesity in children is a decrease in physical activity level and an increase in sedentary lifestyle. Even though approximately 61% of children ages 3 - 5 years of age spend a part of their day in some form of early child care program (day care centers, nursery schools, Head Start, and pre-kindergarten programs) only a few studies have been conducted to examine their daily physical activity level while they are attending preschool. Since the majority of young children spend a part of their day in a preschool setting, this setting could potential play an integral role in increasing their daily physical activity level.

Experts have recommended that in order to meet the current guidelines for daily physical activity (at least 120 minutes/day), planned and/or free playtime should be incorporated into a preschooler's daily schedule. Direct observation indicates that preschoolers spend 27 - 40% of their recess time engaged in moderate-to-vigorous physical activity. By increasing children's time in recess it is possible to increase their daily physical activity level. Therefore the purpose of this study is to examine the effects of increasing the amount of time spent in recess on overall daily physical activity in preschool age children.

Following preliminary screening, participants selected to participant in this study will undergo baseline assessment. All participants will complete two days of baseline conditioning prior to the initiation of the experimental intervention. The experimental intervention will consist of adding an additional recess period for two consecutive school days. Participants' physical activity will be monitored during the baseline conditioning and intervention days. The experimental intervention will last for one week.

ELIGIBILITY:
Inclusion Criteria:

- Hispanic children between 3 - 5 years of age on the date of randomization. A child is defined as Hispanic if their parent/guardian identifies the child's ethnicity as "Hispanic" or "Latino", regardless of race.

Exclusion Criteria:

Children will not be eligible if they have a condition limiting their participation in the intervention (unable to participate in routine outdoor play time at school, requiring oxygen supplementation for exertion, developmental or physical disability preventing participations in the interventions, participants who can not increase their physical activity for any reason); if they have a condition limiting participation in the assessment (parent/guardian is not able to read surveys in English or Spanish, if child is unable to wear the activity monitor); or if parent/guardian is unable to read, understand or complete informed consent in English or Spanish.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60
Dates: Start 2005-12; Study Completion 2006-03

PRIMARY OUTCOMES:
Children's physical activity levels will be monitored Monday thru Friday of the experimental intervention week using the ActiGraph Accelerometer

CONTACTS AND LOCATIONS:
Overall Officials: Sofiya Alhassan, Ph.D., Principal Investigator — Stanford University
Locations (1):
- Roosevelt Elementary School, Redwood City, California, United States